CLINICAL TRIAL: NCT04036019
Title: A Study Evaluating Safety and Efficacy of CBM.CD20 CAR-T(C-CAR066) in Subjects With r/r B Cell Lymphoma Who Received CD19 CAR-T Therapy
Brief Title: A Study of C-CAR066 in Subjects With r/r B Cell Lymphoma Who Received CD19 CAR-T Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Collaborators: Shanghai AbelZeta Ltd. (Industry)
Responsible Party: Principal Investigator, Aibin Liang，MD，Ph.D., Director，Department of Hematology, Shanghai Tongji Hospital, Tongji University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0504-009
Record Dates: First submitted 2019-07-08; First posted 2019-07-29 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: B Cell Lymphoma
Keywords: B cell lymphoma received prior CD19 CAR-T therapy
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-CAR066 (Experimental): Autologous C-CAR066 (CD20-directed CAR T-cell) administered by intravenous (IV) infusion
  Interventions: Biological: CD20-directed CAR-T cells with CliniMACS Prodigy® system

INTERVENTIONS:
Biological: CD20-directed CAR-T cells with CliniMACS Prodigy® system — Autologous 2nd generation CD20-directed CAR-T cells, single infusion intravenously
  Other Names: C-CAR066

SUMMARY:
This is a single-center, non-randomized clinical study to evaluate the safety and efficacy of C-CAR066 in treatment of r/r B cell lymphoma who received CD19 CAR-T therapy.

DETAILED DESCRIPTION:
This study plans to enroll 10 patients to assess the safety and efficacy of C-CAR066. Subjects who meet the eligibility criteria will receive a single dose of C-CAR066 injection.

The study will include the following sequential phases: Screening, Pre- Treatment (Cell Product Preparation, Lymphodepleting Chemotherapy), C-CAR066 infusion and Follow-up Visit.

ELIGIBILITY:
Inclusion Criteria:

1. The patient volunteered to participate in the study, and signed the Informed Consent
2. Age 18-70 years old, male or female
3. Patients with CD20+ DLBCL (including PMBCL and tFL), FL and MCL, at least one measurable lesion (LDi≥ 1.5 cm)
4. r/r lymphoma patients who received prior CD19 CAR-T therapy
5. At least one week from last treatment (radiation, chemotherapy, mAb, etc) to apheresis
6. No immunosuppressive therapy was used within 1 week before C-CAR066 infusion
7. No mAb treatment within 2 weeks before C-CAR066 infusion
8. Adequate organ and bone marrow function
9. No contraindications of apheresis
10. Expected survival time > 3 months
11. ECOG scores 0-1

Exclusion Criteria:

1. Have a history of allergy to cellular products
2. Patients with cardiac insufficiency classified as Class III or IV according to the New York Heart Association (NYHA) Heart Function Classification Standard
3. A history of craniocerebral trauma, consciousness disorder, epilepsy, cerebral ischemia or hemorrhagic cerebrovascular disease
4. Patients with active CNS involvement
5. Patients with autoimmune disease, immunodeficiency, or other treatment requiring immunosuppressor
6. Severe active infection (except simple urinary tract, bacterial pharyngitis), or currently receiving intravenous antibiotics. However, prophylactic antibiotics, antiviral and antifungal treatments are allowed
7. Live vaccination within 4 weeks before apheresis
8. HIV, HBV, HCV and TPPA / RPR infections, and HBV carriers
9. Have a history of alcoholism, drug addiction and mental illness
10. Non-sterile subjects had any of the following: a) being pregnant / lactating; or b) having a pregnancy plan during the trial; or c) having fertility without taking effective contraception
11. Patients with severe fludarabine or cyclophosphamide hypersensitivity
12. The patient has a history of other primary cancers, except for the following:

    1. Non-melanoma such as skin basal cell carcinoma cured by resection
    2. Cured carcinoma in situ such as cervical, bladder or breast cancer
13. The investigators believe that there are other circumstances that are not suitable for the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 12 weeks after C-CAR066 infusion
  The incidence of treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 24 months after C-CAR066 infusion
  The percentage of subjects who achieved complete response and partial response
Complete response rate (CRR) | Up to 24 months after C-CAR066 infusion
  The percentage of subjects who achieved complete response
Duration of response (DOR) | Up to 24 months after C-CAR066 infusion
  The time from the date of first response (PR or CR) to the date of disease progression or death after C-CAR066 infusion
Progression free survival (PFS) | Up to 24 months after C-CAR066 infusion
  The time from C-CAR066 infusion to the date of progression as assessed by Lugano 2014 criteria or death
Overall survival (OS) | Up to 24 months after C-CAR066 infusion
  Time from C-CAR066 infusion to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Aibin Liang, MD,Ph.D., Principal Investigator — Shanghai Tongji Hospital, Tongji University School of Medicine
Locations (1):
- Shanghai Tongji Hospital, Tongji University School of Medicine, Shanghai, China

REFERENCES:
- [Derived] Li P, Liu W, Zhou L, Ye S, Zhu D, Huang J, Li J, Zheng C, Zhu S, Yao X, Zhu K, Yao Y, Qiu L, Liang A, Zou D. C-CAR066, a novel fully human anti-CD20 CAR-T therapy for relapsed or refractory large B-cell lymphoma after failure of anti-CD19 CAR-T therapy: A phase I clinical study. Am J Hematol. 2024 Dec;99(12):2306-2312. doi: 10.1002/ajh.27488. Epub 2024 Oct 1. PMID 39351902